CLINICAL TRIAL: NCT07373795
Title: Gummy Candies Containing Maqui Berry (Aristotelia Chilensis) to Improve Glycemic Control of Overweight Subjects
Brief Title: Gummy Candies With Maqui Berry
Acronym: MaquiGUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonzalo Jorquera, PhD (Other)
Collaborators: Universidad de Valparaiso (Other)
Responsible Party: Sponsor-Investigator, Gonzalo Jorquera, PhD, Assistant professor, University of Chile
Organization: University of Chile (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DIUV-CIDI 15/2024; 100-InES/Lánzate-UV 2022 (Other: University of Valparaíso)
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Overweight (BMI > 25); Obesity & Overweight; Insulin Resistance Syndrome; Type 2 Diabetes
Keywords: Maqui berry; GLP-1; Polyphenols; glycemic control; Antioxidant response; SOD; Catalase; TRAP
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Intervention Participants will complete a three-condition, within-subject acute intervention with one-week washouts between visits: (i) baseline/control: 150 g white bread (75 g available carbohydrate); (ii) white bread + GM: 150 g white bread plus 24 g GM (3 gummies); and (iii) white bread + GMM: 150 g white bread plus 24 g GMM (3 gummies). Each participant will serve as their own control. On each study day (control, GM, GMM), a fasting baseline sample (time 0) will drawn before ingestion of the test meal. Visits will occur on separate days, one week apart, under standardized pre-test conditions (overnight fast, fixed morning schedule, and pre specified diet/activity restrictions).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control, GM, GMM (Other): Participants will complete a three-condition, within-subject acute intervention with one-week washouts between visits: (i) baseline/control: 150 g white bread (75 g available carbohydrate);(ii) white bread + GM: 150 g white bread plus 24 g GM (3 gummies); (iii) white bread + GMM: 150 g white bread plus 24 g GMM (3 gummies). Each participant will serve as their own control. On each study day (control, GM, GMM), a fasting baseline sample (time 0) will drawn before ingestion of the test meal. Visits will occur on separate days, one week apart, under standardized pre-test conditions (overnight fast, fixed morning schedule, and pre specified diet/activity restrictions).
  Interventions: Dietary Supplement: GM; Dietary Supplement: Control; Dietary Supplement: GMM

INTERVENTIONS:
Dietary Supplement: GM — white bread + GM: 150 g white bread plus 24 g GM (3 gummies)
Dietary Supplement: Control — Baseline/control: 150 g white bread (75 g available carbohydrate)
Dietary Supplement: GMM — white bread + GM: 150 g white bread plus 24 g GM (3 gummies)

SUMMARY:
The goal of this clinical trial is to learn if Maqui berry gummy encapsulated (GMM) compared to non-encapsulated (GM) can improve glycemic response in overweight adults. It will also learn about the possible effect of serum antioxidant levels. The main questions it aims to answer are:

Does GMM or GM low the glycemic response in overweight/obese subjects after consuming a carbohydrate rich food?

Does GMM or GM increase antioxidant levels in overweight/obese subjects after consuming a carbohydrate rich food?

Researchers will compare (i) a carbohydrate rich food, (ii) GMM + a carbohydrate rich food, (iii) GM + a carbohydrate rich food to see if Maqui gummy work to control glycemic and antioxidant levels.

Participants will:

Take a carbohydrate rich food, and/or Maqui gummy three times, one week apart Have blood samples collected and answer food questionnaires in each visit

DETAILED DESCRIPTION:
Inclusion and exclusion criteria for intervention Ten sedentary volunteers will be recruited. Inclusion criteria: body mass index (BMI) of overweight or obesity (BMI at least 25.0 kg/m2); absence of non-communicable chronic disease; and sedentary (less than 30 minutes of physical activity for 3 times a week). All participants will be asked to maintain their physical activity, food intake and medications during the whole study. Exclusion criteria: use of hypoglycemic drugs, supplements containing antioxidants, and high consumption of polyphenols (more than 2 g per day); food allergy to Maqui berry or any component from the GCs; pregnancy or lactation. The study was approved by the Ethics Committee of the Faculty of Pharmacy, Universidad de Valparaíso (CBI 014/2022).

Participant characteristics Weight and height will be determined to calculate BMI, as well as waist circumference and triceps fold. Food Frequency Questionnaires (FFQ) will be recovered prior to the study to estimate fiber and total dietary antioxidant intake, mainly polyphenols, carotenes, and vitamin E and C consumption. All intervention was performed on the Faculty of Pharmacy, Universidad de Valparaíso, by capacity personal.

Intervention Participants will complete a three-condition, within-subject acute intervention with one-week washouts between visits: (i) baseline/control: 150 g white bread (75 g available carbohydrate); (ii) white bread + GM: 150 g white bread plus 24 g GM (3 gummies); and (iii) white bread + GMM: 150 g white bread plus 24 g GMM (3 gummies). Each participant will serve as their own control. On each study day (control, GM, GMM), a fasting baseline sample (time 0) will drawn before ingestion of the test meal. Visits will occurr on separate days, one week apart, under standardized pre-test conditions (overnight fast, fixed morning schedule, and prespecified diet/activity restrictions).

Control condition and mitigation of expectancy bias Our control condition will use the white-bread-only day served as the no-Maqui control for glycemic and antioxidant responses. Interventions will add 24 g of gummies (3 units) to the same bread load. The investigators will not include a separate "placebo gummy" because the study is a pilot designed around an objective white-bread control, and producing a sensorially indistinguishable polyphenol-free gummy is challenging (Maqui pigments/flavor); even GM vs. GMM differed in smell and taste in our sensory testing, suggesting blinding with a placebo matrix would likely be imperfect. To limit expectancy effects and mitigate possible bias, the investigators: (i) will use objective endpoints (glycemia/insulin/GLP-1; TRAP, SOD, CAT); (ii) enforce standardized pre-test conditions (12 h fast; morning testing at fixed hours; dietary/activity restrictions with documented adherence); and (iii) implement one-week washouts between interventions. All comparisons will be within-person relative to the white-bread control.

Blood sample procedures Blood samples will be collected from the participants after a 12 h overnight fast at the beginning of each intervention and during a 2 h period. Samples will be collected in sodium heparin tubes (final concentration of 0.1%). For insulin and GLP-1 determinations, blood will be centrifuged at 2000× g for 10 minutes at 4 ◦C and the supernatant will be frozen at -80 ◦C. For the antioxidant status measurements, plasma will be separated from the red cells via centrifugation at 1500× g for 1 min at 4 ◦C. Plasma will be immediately frozen at -80 ◦C for subsequent total reactive antioxidant power (TRAP) analysis, while red cells will be washed with bovine serum albumin (BSA), centrifuge 3 times at 1500× g for 15 minutes, discarding the supernatant each time. Before storage at -80°C, the red cells will be diluted with a hypotonic solution for catalase (CAT, ratio 1:10) and superoxide dismutase (SOD, ratio 1:28) for further analysis.

Antioxidant status biomarkers Total Reactive Antioxidant Power (TRAP) Briefly, 10 µL of supernatant will be mix with a 1:1 mixture of 150 µM 2,20-azino-bis(3-ethylbenzothiazoline-6-sulfonic acid) and 10 mM 2,20-azobis(2-amidinopropane), previously incubate at 45 °C during 30 minutes. Kinetics will determine at 734 nm for 10, 30, and 50 seconds after adding the sample. The antioxidant capacity will be measure comparing to Trolox®.

Total protein measurement Total protein quantification will be performed using erythrocytes to normalize SOD and CAT enzyme activity. For this, the Pierce BCA Protein Assay Kit (Thermofisher) will be used, based on an albumin curve made from an Albumin Standart (Thermofisher). All protocols will be used according to the manufacturer.

Superoxide dismutase (SOD) This assay is based on the reduction of cytochrome c by the superoxide radical in a xanthine/xanthine oxidase system. Briefly, 5 µL of homogenized samples will be mixed with 0.5 mM xanthine (Sigma-Aldrich, St. Louis, MO, USA) and 20 µM cytochrome C (Sigma-Aldrich, St. Louis, MO, USA) dissolved in a phosphate buffer. This solution will be mixed with xanthine oxidase (Sigma-Aldrich, St. Louis, MO, USA) and 0.1 mM EDTA (1:40). Enzymatic activity will be detected at 550 nm in a Rayleigh UV-2601 spectrophotometer. Each sample will be analyzed in triplicate.

Catalase (CAT) The catalase activity will be determined by measuring the loss of absorbance at 240 nm of a reaction mixture consisting of 100 µL of 0.3 M H2O2 (Merck, Darmstadt, Germany) in 2.9 mL of phosphate buffer (50 mM Na2HPO4 and 50 mM NaH2PO4, pH 7.8) and 50 µL of samples. Measurements will be performed during 90 seconds in a Rayleigh UV-2601 spectrophotometer. Each sample will be analyzed in triplicate.

Glucose, Insulin and GLP-1 Blood capillary samples will be obtained from participant's finger using glucose test strips (One Touch II) before consuming the white bread (time 0) and after consumption with or without the gummies (at 15, 30, 60, 90 and 120 minutes). Blood samples will be obtained for insulin concentrations at time points 0 and 120 minutes, that will be measured using a chemiluminescence immunoassay according manufacturer's recommendations. Human plasma levels of GLP-1 will be measure at 0 and 120 minutes using the GLP-1 ELISA Kit (BMS2194; ThermoFisher Cientific) following the manufacturer's instructions. The incremental area under the curve (AUC) each 120 minutes of plasma glucose, insulin and GLP-1 will be calculated by using trapezoidal rule with fasting values considered as baseline.

Statistical analysis Sample size and power: This study will conceived as an early-phase, acute, within-subject intervention in which each participant served as their own control across three conditions (baseline, GMM, GM) with a one-week washout. Given the efficiency of within-subject designs, investigators are planning a modest sample size (n = 10 completers). A sensitivity analysis indicates that, for two-sided paired comparisons with α = 0.05 and 80% power, n = 10 can detect a large standardized within-subject effect of approximately Cohen's dz ≈ 0.9-1.0. Shapiro-Wilk test will be used to confirm normality of the data. Spearman's rank correlations will be used within each intervention condition (analyzing GM and GMM separately) to examine associations between postprandial glycemic, insulinemic and GLP-1 exposures (glycemic AUC, insulin AUC and GLP-1 AUC), and antioxidant-related variables: SOD activity, plasma TRAP (TEAC), catalase activity, and dietary intakes from the FFQ (vitamin C, vitamin E, carotenes, total polyphenols, and fiber). Investigators will report Spearman coefficient and two-sided p-values (n = 10). Given the pilot, hypothesis-generating nature of the study, analyses will be exploratory and do not imply causality; multiplicity adjustments will not be applied. Multiple comparisons will made using Kruskal-Wallis test assuming the p value of less than 0.05 as significant. All analysis will be performed with GraphPad Prism software version 9.0.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of overweight or obesity (BMI at least 25.0 kg/m2);
* absence of non-communicable chronic disease;
* being sedentary (less than 30 minutes of physical activity for 3 times a week).
* All participants must maintain their physical activity, food intake and medications during the whole study.

Exclusion Criteria:

* use of hypoglycemic drugs
* supplements containing antioxidants
* high consumption of polyphenols (more than 2 g per day)
* food allergy to Maqui berry or any component from the GCs
* pregnancy or lactation in the case of the female participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Glycemia | Blood capillary samples will be obtained from participant's finger using glucose test strips (One Touch II) before consuming the white bread (time 0) and after consumption with or without the GCs (at 15, 30, 60, 90 and 120 minutes).
  Blood capillary samples were obtained from participants' fingers using glucose test strips (One Touch II) before consuming the white bread (time 0) and after consumption with or without the GCs (at 15, 30, 60, 90 and 120 minutes). It will be expressed as mg/dl.

SECONDARY OUTCOMES:
Insulin levels | Blood samples will be obtained for insulin concentrations at time points 0 and 120 minutes that will be measured using a chemiluminescence immunoassay according manufacturer's recommendations.
  Insulin AUC: Blood samples will be obtained for insulin concentrations at time points 0 and 120 minutes, which will be measured using a chemiluminescence immunoassay according to the manufacturer's recommendations. It will be expressed as mg/dl.
GLP-1 | Human plasma levels of GLP-1 will be measured at 0 and 120 minutes.
  Human plasma levels of GLP-1 will be measured using the GLP-1 ELISA Kit (BMS2194; ThermoFisher Cientific) following the manufacturer's instructions. The incremental area under the curve (AUC) each 120 minutes of GLP-1 will be calculated by using trapezoidal rule with fasting values considered as baseline. It will be expressed as mg/dl.
Total Reactive Antioxidant Power (TRAP) | Antioxidant biomarkers will be measured at 0 and 120 minutes after each intervention
  Briefly, 10 µL of supernatant will be mixed with a 1:1 mixture of 150 µM 2,20-azino-bis(3-ethylbenzothiazoline-6-sulfonic acid) and 10 mM 2,20-azobis(2-amidinopropane), previously incubated at 45 °C during 30 minutes. Kinetics will be determined at 734 nm for 10, 30, and 50 seconds after adding the sample. Antioxidant capacity will be measured compared to Trolox®. The results will be expressed as micromolar of Trolox® equivalent antioxidant capacity (µM TEAC).
Total protein measurement | Antioxidant biomarkers will be measured at 0 and 120 minutes after each intervention
  Total protein quantification will be performed using erythrocytes to normalize SOD and CAT enzyme activity. For this, the Pierce BCA Protein Assay Kit (Thermo Fisher) will be used, based on an albumin curve made from an Albumin Standard (Thermo Fisher). All protocols will be used according to the manufacturer. It will be expressed as mcg/dl.
Superoxide dismutase (SOD) | Antioxidant biomarkers will be measured at 0 and 120 minutes after each intervention
  Briefly, 5 µL of homogenized samples will be mixed with 0.5 mM xanthine (Sigma-Aldrich, St. Louis, MO, USA) and 20 µM cytochrome c (Sigma-Aldrich, St. Louis, MO, USA) dissolved in a phosphate buffer. This solution will be mixed with xanthine oxidase (Sigma-Aldrich, St. Louis, MO, USA) and 0.1 mM EDTA (1:40). Enzymatic activity will be detected at 550 nm in a Rayleigh UV-2601 spectrophotometer. Each sample will be analyzed in triplicate. Results will be expressed as units of enzyme per microgram of protein (UE/µg protein).
Catalase (CAT) | Antioxidant biomarkers will be measured at 0 and 120 minutes after each intervention.
  The catalase activity will be determined by measuring the loss of absorbance at 240 nm of a reaction mixture consisting of 100 µL of 0.3 M H2O2 (Merck, Darmstadt, Germany) in 2.9 mL of phosphate buffer (50 mM Na2HPO4 and 50 mM NaH2PO4, pH 7.8) and 50 µL of sample. Measurements will be performed for 90 seconds in a Rayleigh UV-2601 spectrophotometer. Each sample will be analyzed in triplicate. Results will be expressed as units of enzyme per micrograms of protein (UE/µg protein).
Waist circumference | At the beginning
  It will be measure with metric. It will be expressed as cm.
Food Frequency Questionnaires (FFQ) | At the beginning
  Food Frequency Questionnaires (FFQ) will be collected prior to the study to estimate fiber and total dietary antioxidant intake, mainly polyphenols, carotenes, and vitamin E and C consumption. FFQ analyses will be based on the Chilean Food Composition Table and the USDA National Nutrient Database for Standard Reference. It will be expressed as mg/day of consumption.

OTHER OUTCOMES:
IMC | At the beginning
  Weight (kg) and height (cm) will be determined to calculate BMI (kg/cm2)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Valparaíso, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided